CLINICAL TRIAL: NCT03080948
Title: Cutaneous Melanoma Risk Stratification of Individuals With a High-Risk Nevus Phenotype
Brief Title: Risk Stratification Among Individuals Who Have Many Moles on Their Skin
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Princess Alexandra Hospital, Brisbane, Australia (Other); Sheba Medical Center (Other Government); Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 17-083
Record Dates: First submitted 2017-03-10; First posted 2017-03-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: High-Risk Nevus Phenotype
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- History of Melanoma (cases): Participants at high-risk for melanoma (that is, those having many nevi and morphologically atypical nevi) who either have a history of invasive melanoma (cases) or do not have a history of melanoma (controls) and will perform comprehensive total body imaging of their moles in order to identify phenotypic markers of melanoma risk that aid in melanoma risk stratification. In addition, we will investigate histopathologic and molecular features of moles that are associated with melanoma risk and with melanoma subtypes. The evaluations needed for this study protocol will be primarily performed during routine clinical care.
  Interventions: Behavioral: survey; Other: Saliva samples
- No Melanoma History (controls): Participants at high-risk for melanoma (that is, those having many nevi and morphologically atypical nevi) who either have a history of invasive melanoma (cases) or do not have a history of melanoma (controls) and will perform comprehensive total body imaging of their moles in order to identify phenotypic markers of melanoma risk that aid in melanoma risk stratification. In addition, we will investigate histopathologic and molecular features of moles that are associated with melanoma risk and with melanoma subtypes. The evaluations needed for this study protocol will be primarily performed during routine clinical care.
  Interventions: Behavioral: survey; Other: Saliva samples

INTERVENTIONS:
Behavioral: survey — Research assessments as part of this protocol will be scheduled during routine clinic visits
Other: Saliva samples — Germline DNA analysis

SUMMARY:
The investigators are doing this study to improve our ability to identify which people with many moles on their skin are most likely to develop skin melanoma. The investigators hope to identify features of moles that are associated with melanoma risk. The investigators hope to use this information to customize and tailor melanoma screening to the individual patient based on a better estimate of their individual risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* High-risk nevus phenotype (≥ 50 nevi (≥ 2mm in size) and ≥ 1 atypical nevus)
* First presented to MSKCC for cutaneous melanoma-related care on or after April 2016
* Cases: diagnoses of unequivocal invasive cutaneous melanomas (AJCC Stages I-IV) confirmed by MSKCC pathology on or after April 2016
* Cases: completion of surgical treatment of primary melanoma
* Ability to sign or verbally consent to the informed consent

Exclusion Criteria:

* Controls: Histopathologically borderline melanocytic tumors for which melanoma could not be excluded or that were treated as possible melanomas.
* Known germline high-penetrance melanoma predisposition mutation (that is, CDKN2A, CDK4, and BAP1)
* Cases: history of invasive cutaneous melanoma (AJCC Stages I-IV) not confirmed by MSKCC pathology
* History of acrolentiginous type of cutaneous melanoma or history of mucosal melanoma
* Cases and controls: prior administration of systemic medications known to modify nevus phenotype, including but not limited to: MEK inhibitors (trametinib, cobimetinib, etc.), BRAF inhibitors (vemurafenib, dabrafenib, etc.), and immunotherapy (pembrolizumab, nivolumab, atezolizumab, ipilimumab, etc.). Controls: history of Stage 0-IV melanoma confirmed by MSKCC pathology
* History of limb amputation or other condition (e.g., tattoos, burns) per investigator discretion that would modify nevus phenotype
* Physical inability to undergo total body photography or reflectance confocal microscopy imaging (that is, remain relatively still for durations of 3-5 minutes)
* Known hypersensitivity to adhesive rings used for reflectance confocal microscopy
* Inability to give informed consent
* Have skin afflicted with anther skin condition (for example, psoriasis) that would affect ability to characterize nevus phenotype (per investigator discretion)
* Familial cutaneous melanoma history (families with at least one invasive melanoma and two or more other diagnoses of invasive melanoma or pancreatic cancer among first- or second-degree relatives on the same side of the family). We will confirm melanoma family history via medical record documentation, whenever possible, as recommended by previous studies that disproved about half of the reported family histories of melanoma among first-degree relatives in case-control studies.
* Age 70 or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the Melanoma Screening and Surveillance Program (MSSP).
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
number of patients having specific dermoscopic patterns | 2 years
  For each person, the proportions of their nevi having specific dermoscopic patterns will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Halpern, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center Hauppauge, Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm